CLINICAL TRIAL: NCT05181150
Title: Gut Peptides and Bone Remodeling in Individuals With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kirsa Skov-Jeppesen, Principal investigator, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CBC-SCI-21
Record Dates: First submitted 2021-12-18; First posted 2022-01-06 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injury; GIP; GLP-2; CTX; P1NP; Bone resorption; Bone formation; Bone turnover; Bone remodeling
MeSH Terms: conditions — Spinal Cord Injuries; Bone Resorption

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Meal test (Experimental)
  Interventions: Other: Meal test
- GIP, Glucose-dependent insulinotropic polypeptide (Experimental)
  Interventions: Other: GIP
- GLP-2, Glucagon-like-peptide-2 (Experimental)
  Interventions: Other: GLP-2
- GIP + GLP-2 (Experimental)
  Interventions: Other: GIP + GLP-2
- Placebo (saline) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Meal test — Ingestion of an oral liquid meal (nutridrink), 200 mL.
  Other Names: Nutridrink
  Arms: Meal test
Other: GIP — Subcutaneous GIP injection.
  Arms: GIP, Glucose-dependent insulinotropic polypeptide
Other: GLP-2 — Subcutaneous GLP-2 injection.
  Arms: GLP-2, Glucagon-like-peptide-2
Other: GIP + GLP-2 — Subcutaneous GIP + GLP-2 injection.
  Arms: GIP + GLP-2
Other: Placebo — Subcutaneous saline injection.
  Arms: Placebo (saline)

SUMMARY:
Both GLP-2 and GIP reduce bone resorption (measured as CTX) in healthy persons. In this study, we will investigate whether GLP-2 and GIP is reducing CTX in individuals with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria (Individuals with spinal cord injury):

* Spinal cord injury resulting in the need of a wheelchair
* BMI: 16-32 kg/m2

Inclusion Criteria (Healthy controls):

* Intact spinal cord
* Matched on gender, age and BMI to the group with spinal cord injury

Exclusion Criteria:

* Treatment with antidiabetics
* Treatment with anti-resorptive agents
* Gastrointestinal disease
* Smoking
* Long term steroid treatment
* Weight change more than 3 kg within the last 3 months.
* Overweight or intestinal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
CTX | -10 to 240 minutes
  Bone resorption measured as collagen type 1 C-terminal telopeptide (CTX) in serum.

SECONDARY OUTCOMES:
P1NP | -10 to 240 minutes
  Bone formation measured as procollagen type 1 N-terminal propeptide (P1NP) in serum.
PTH | -10 to 240 minutes
  PTH measured in serum PTH measured in serum
Sclerostin | -10 to 240 minutes
  Bone marker
Glucose | -10 to 240 minutes
  Measured in serum
Insulin | -10 to 240 minutes
  Measured in serum
C-peptide | -10 to 240 minutes
  Measured in serum
GIP | -10 to 240 minutes
  Glucose-dependent insulinotropic polypeptide measured in plasma
GLP-2 | -10 to 240 minutes
  Glucagon-like peptide 2 measured in plasma.
Glucagon | -10 to 240 minutes
  Glucagon measured in plasma
Blood pressure | -10 to 240 minutes
  Measured before blood sampling
Heart rate | -10 to 240 minutes
  Measured before blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Mette M Rosenkilde, Prof., MD, Study Director — University of Copenhagen
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No